CLINICAL TRIAL: NCT04106427
Title: Brain Stimulation And Group Therapy to Improve Gesture and Social Skills in Psychosis (BrAGG-SoS) - a Randomized, Placebo-controlled, Double-blind Trial of Transcranial Magnetic Stimulation and Group Therapy
Brief Title: Brain Stimulation And Group Therapy to Improve Gesture and Social Skills in Psychosis (BrAGG-SoS)
Acronym: BrAGG-SoS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-00798
Record Dates: First submitted 2019-09-17; First posted 2019-09-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia
Keywords: gesture; rTMS; cognitive remediation; social cognitive remediation therapy
MeSH Terms: conditions — Schizophrenia; Gestures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Assessments will be conducted by blind assessors. Participants will be blind to the type of psychotherapy and the type of rTMS administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cTBS plus SCRT (Experimental): 10 daily sessions of continous theta burst (cTBS) on the right inferior parietal cortex for two weeks together with 16 sessions of social cognitive remediation therapy (SCRT) twice per week over an eight week period according to the manual
  Interventions: Device: continuous theta burst stimulation (cTBS); Behavioral: social cognitive remediation therapy (SCRT)
- Placebo plus SCRT (Placebo Comparator): 10 daily sessions of placebo continous theta burst (cTBS) on the right inferior parietal cortex for two weeks together with 16 sessions of social cognitive remediation therapy (SCRT) twice per week over an eight week period according to the manual
  Interventions: Device: placebo cTBS; Behavioral: social cognitive remediation therapy (SCRT)
- Sham SCRT (Sham Comparator): 16 sessions of sham social cognitive remediation therapy (SCRT) twice per week over an eight week period. Participants will engage in non-effective group activities
  Interventions: Behavioral: Sham group therapy

INTERVENTIONS:
Device: continuous theta burst stimulation (cTBS) — cTBS stimulation of 17 mins over right inferior parietal lobe (IPL) with two 44 s stimulations separated by 15 mins, 10 sessions in total (5 per week). intensity will be 100% of resting motor threshold at 30 Hz.
  administered in weeks 1 and 2 of the trial
  Arms: cTBS plus SCRT
Device: placebo cTBS — Placebo stimulation of 17 mins over right IPL with two 44 s stimulations separated by 15 mins, 10 sessions in total (5 per week). intensity will be 0% of resting motor threshold at 30 Hz.
  administered in weeks 1 and 2 of the trial
  Arms: Placebo plus SCRT
Behavioral: social cognitive remediation therapy (SCRT) — 16 sessions of group SCRT will be scheduled within 8 weeks, comprising 6-8 participants per group with 2 therapists. Duration of group sessions will be 60-90 mins. The content will follow the manual of SCRT and we will add a short intervention to practice the use of co-speech gestures at each session
  Arms: Placebo plus SCRT; cTBS plus SCRT
Behavioral: Sham group therapy — Group activities in closed groups of 6 participants. Schedule of two sessions per week for 8 weeks. Two therapists are guiding different leisure activities, e.g. group walks, going to museums/movies, games.
  Arms: Sham SCRT

SUMMARY:
Randomized, double-blind, placebo-controlled clinical trial testing the effects of 10 sessions of continuous theta burst stimulation and the effects of 16 sessions of social cognitive remediation therapy on gesture performance and nonverbal communication skills in schizophrenia

DETAILED DESCRIPTION:
The study focuses on nonverbal communication skills in schizophrenia. The trial will test, whether the combination of noninvasive brain stimulation and group psychotherapy will improve gesture performance and thus nonverbal communication in schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Right-handed subjects
* Ability and willingness to participate in the study
* Ability to provide written informed consent
* Informed Consent as documented by signature
* schizophrenia spectrum disorders according to Diagnostic and statistical manual version 5 (DSM-5)

Exclusion Criteria:

* Substance abuse or dependence other than nicotine
* Past or current medical or neurological condition associated with impaired or aberrant movement, such as brain tumors, stroke, M. Parkinson, M. Huntington, dystonia, or severe head trauma with subsequent loss of consciousness.
* Epilepsy or other convulsions
* History of any hearing problems or ringing in the ears
* Standard exclusion criteria for cerebral magnetic resonance imaging scanning and transcranial magnetic stimulation (TMS); e.g. metal implants, claustrophobia
* Patients only: any transcranial magnetic stimulation (TMS) treatment in the past 3 months
* Patients only: any cognitive remediation therapy in the past 2 years
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
change in gesture performance using the Test of Upper Limb Apraxia (TULIA) | baseline, week 2, week 8, week 32
  Test of upper limb apraxia (TULIA), recorded on video and scored according to manual. contains 48 items (gestures performed on verbal or visual instruction), total score ranges 0-240; higher scores indicate better performance.

SECONDARY OUTCOMES:
change in the profile of nonverbal sensitivity (PONS) | baseline, week 2, week 8, week 32
  profile of nonverbal sensitivity (PONS), short test of the interpretation of video clips, total score will be evaluated, higher scores indicate better performance
change in Brief Negative Symptoms Scale (BNSS) | baseline, week 2, week 8, week 32
  rating instrument to assess severity of negative symptoms with 13 items, total score will be used ranging 0-78, higher scores indicate higher symptom severity
change in Self evaluation of negative symptoms (SNS) | baseline, week 2, week 8, week 32
  questionnaire on subjective negative symptoms, includes 20 items. total scores will be used ranging 0-40 with higher scores indicating increased symptom severity
change in Social and occupational functioning (SOFAS) | baseline, week 2, week 8, week 32
  rating scale on community functioning, total score is used ranging 0-100, higher scores indicated better functioning
change in the specific level of functioning assessment scale (SLOF) | baseline, week 2, week 8, week 32
  rating scale on community functioning, total scores are used ranging 43-215 with higher scores indicating better functioning
change in functional capacity (UPSA brief) | baseline, week 2, week 8, week 32
  brief version of the University of California in San Diego Performance-based Skills Assessment (UPSA-brief), short assessment of skills, total scores are used ranging from 0-100 with higher scores indicating better skill performance
change in neural activity during gesture planning using functional magnetic resonance imaging (fMRI) | baseline, week 8
  pantomime task during functional magnetic resonance imaging. Blood oxygenation level depended (BOLD) signal change from baseline to week 8 will be compared during gesture planning within the cerebral praxis network. Standard fMRI analyses procedures will be applied
number of participants with treatment related adverse events as assessed with rating scale | week 2
  after each repetitive transcranial magnetic stimulation (rTMS) session participants will be inquired about adverse events. after 5 sessions and after 10 sessions, a structured questionnaire will be applied following the guidelines for rTMS treatment. This will assess specific adverse events and their severity

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Walther, MD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Translational Research Center, University Hospital of Psychiatry, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chapellier V, Pavlidou A, Mueller DR, Walther S. Brain Stimulation and Group Therapy to Improve Gesture and Social Skills in Schizophrenia-The Study Protocol of a Randomized, Sham-Controlled, Three-Arm, Double-Blind Trial. Front Psychiatry. 2022 Jul 7;13:909703. doi: 10.3389/fpsyt.2022.909703. eCollection 2022. PMID 35873264